CLINICAL TRIAL: NCT02498873
Title: Linear Running Periodization x Nonlinear: a Cross Effect of Five Months Controlled Running on VO2Max and Critical Power Performance
Brief Title: Linear Running Periodization x Nonlinear
Acronym: Running
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Alberto Souza de Sá Filho, Doctorade in Mental Health, Universidade Federal do Rio de Janeiro
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UNIVERSO-01
Record Dates: First submitted 2015-07-11; First posted 2015-07-15 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: VO2Max; Physical Conditioning; Aerobic Exercise; Performance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Linear Periodization (Active Comparator): Linear Periodization Running (Crossover Design)
  Interventions: Behavioral: Non Linear Periodization
- Non Linear Periodization (Active Comparator): Non Linear Periodization Running (Crossover Design)
  Interventions: Behavioral: Linear Periodization

INTERVENTIONS:
Behavioral: Linear Periodization — Linear Intensity Periodization Running
  Other Names: LP; Progressive Periodization
  Arms: Non Linear Periodization
Behavioral: Non Linear Periodization — Non Linear Periodization Running
  Other Names: NLP; Randomized Intensity
  Arms: Linear Periodization

SUMMARY:
In a competitive scenario, trainers and coaches seek to improve the performance of their athletes organizing macrocycles (year), mesocycles (months), and microcycles (weeks) training aimed at a specific moment of a competition. The organization variables, mainly the intensity of exercise in a training routine can stimulate important physiological pathways and uphold superior gains to VO2max, leading to a peak aerobic performance. However, due to lack of evidence, and the difficulty of control on a large scale, the effects of the intensity organization over a mesocycle periodization are still poorly investigated.

DETAILED DESCRIPTION:
The objective of this study is compare two intensity blocks organization a) linear progression intensity (LP) and b) randomized or not intensity linaer (NLP) over five months running training, and a crossover design between subjects, on gains in VO2max, peak velocity (Vpeak) and critical power (CP). Furthermore, the relationship between the gains obtained with the training and the amount of exercise will be established. In our case all dependent variables will increase after training, with no significant differences between the two strategies on dependent variables.

ELIGIBILITY:
Inclusion Criteria:

* Minimum standards of physical activity proposed by the ACSM
* 18-45 years
* No metabolic or cardiovascular events
* No use ergogenic resources

Exclusion Criteria:

* Sedentary
* Diagnosis of cardiac, pulmonary or diabetes type I or II
* No injuries

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
VO2Max | 0 - 2 month; 1 month (wash out); 3 - 5 month
  Observe the improvement of VO2max

SECONDARY OUTCOMES:
Critical Power | 0 - 2 month; 1 month (wash out); 3 - 5 month
  Performance of Critical Power in Linear Periodization and Non Linear Periodization
Peak Velocity | 0 - 2 month; 1 month (wash out); 3 - 5 month
  Performance of Vpeak in Progressive Effort Test

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio Machado, PhD, Study Director — Universidade Federal do Rio de Janeiro